CLINICAL TRIAL: NCT06583057
Title: Multicenter Comparison of Thermal Ablation Versus Thyroid Lobectomy for Subcapsular Papillary Thyroid Microcarcinoma: a Retrospective Cohort Study
Brief Title: Multicenter Comparison of Thermal Ablation Versus Thyroid Lobectomy for Subcapsular Papillary Thyroid Microcarcinoma
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yukun Luo, Chief of ultrasound, Chinese PLA General Hospital
Other Study IDs: S2019-211-01
Record Dates: First submitted 2024-08-23; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-09

CONDITIONS: Thyroid Cancer; Papillary Thyroid Microcarcinoma
Keywords: Thermal ablation; Lobectomy; Ultrasound; Papillary thyroid microcarcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Papillary Thyroid Microcarcinoma | interventions — Transurethral Resection of Prostate; Ablation Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Thermal ablation group: Patients with clinical T1aN0M0 subcapsular papillary thyroid carcinoma who underwent thermal ablation for treatment.
  Interventions: Procedure: Thermal ablation; Procedure: Thyroid lobectomy
- Thyroid lobectomy group: Patients with clinical T1aN0M0 subcapsular papillary thyroid carcinoma who underwent thyroid lobectomy for treatment.
  Interventions: Procedure: Thermal ablation; Procedure: Thyroid lobectomy

INTERVENTIONS:
Procedure: Thermal ablation — Patients who underwent thermal ablation were performed in the outpatient clinic's operating room under local anesthesia. Thermal ablation was performed under real-time ultrasound-guided. The 18-G bipolar radiofrequency applicator with a 0.9 cm active tip (CelonProSurge micro 100-T09, Olympus Surgical Technologies Europe) , or a 16-G/17-G cooled microwave antenna with a 0.3 cm tip (ECO-100A1, YIGAO MWA system Co., Ltd; KY-2000, Kangyou Medical, Nanjing, China) was used during ablation.
  Other Names: Ablation technique
Procedure: Thyroid lobectomy — Patients who underwent thyroid lobectomy were performed in the operating theater under general anesthesia. Lobectomy (or lobectomy plus isthmusectomy) with prophylactic central neck dissection were performed.

SUMMARY:
To compare the clinical outcomes of Thermal ablation with those of thyroid lobectomy in patients with subcapsular papillary thyroid microcarcinoma.

DETAILED DESCRIPTION:
The global incidence of papillary thyroid microcarcinoma (PTMC) has increased rapidly in recent decades because of improved ultrasound (US) detection and fine needle aspiration biopsy and has primarily contributed to the surge in cases of thyroid carcinoma. Given the indolent characteristics of most PTMCs, the American Thyroid Association guidelines recommend active surveillance for low-risk PTMC to prevent over-treatment. Nevertheless, in many countries, active surveillance poses challenges, including patient anxiety, limited medical resources, and insurance coverage limitations when adopted. Furthermore, many patients prefer treatment rather than active surveillance due to anxiety, a meta-analysis showed that a significant proportion of patients (8.7%-32%) who underwent delayed surgery without tumor progression during active surveillance. Thyroid lobectomy (TL), replacing total thyroidectomy is recommended as the first-line treatment for PTMC by several guidelines. However, there were still concerns remain regarding lifelong hormone replacement therapy, surgery-related complications, and the potential over-treatment associated with TL.

Thermal ablation (TA) has emerged as a viable alternative for the managing of PTMC within the thyroid gland, as evidenced by studies conducted across various Asian and European countries. It has been endorsed as an alternative treatment strategy to TL in clinical guidelines issued by multiple professional associations in Europe, Asia, and North America. However, controversy persists regarding its usefulness for subcapsular PTMC because of concerns about potential extrathyroidal extension (ETE) or occult lymph node metastasis (LNM), which may impact disease progression post-treatment. There are also technical challenges and safety issues when ablating subcapsular lesions. To date, a limited number of studies have reported the short-term efficacy of TA in treating subcapsular PTMC.However, these studies were constrained by small sample sizes and the absence of comparative analyses between the first-line treatment option, TL, and TA. Consequently, further research is needed to fully understand the role of TA in the therapeutic management of subcapsular PTMC and its potential as an alternative to TL.

Therefore, the aim of this multicenter study was to compare the clinical outcomes of TA with those of TL in patients with subcapsular PTMC.

ELIGIBILITY:
Inclusion Criteria:

1. a unifocal papillary thyroid carcinoma (PTC) diagnosed by fine-needle aspiration or core-needle biopsy;
2. tumor with a maximum diameter of ≤ 10 mm detected on ultrasound;
3. tumor located within ≤ 2mm from the thyroid capsule (with or without tumor-associated capsular bulging or capsular discontinuity);
4. absence of clinical or imaging evidence of gross ETE (involvement of strap muscles, obtuse angles between the tumor and trachea/esophagus, protrusion into the tracheoesophageal groove, and invasion into other neck structures);
5. no clinical or imaging evidence suggesting lymph node metastasis or distant metastasis

Exclusion Criteria:

1. aggressive subtypes of PTC (aggressive subtypes of PTC includes the tall cell, columnar cell, solid, and hobnail variants);
2. multifocal PTMC;
3. history of neck surgery or TA;
4. a follow-up period of < 24 months;
5. incomplete follow-up data, or poor-quality pre-treatment ultrasound images

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study included patients with clinical T1aN0M0 PTC who underwent thermal ablation or thyroid lobectomy at three institutions between June 2014 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date of enrollment of the first patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Interval between the date of treatment and the date of detection of disease progression or last follow-up.

SECONDARY OUTCOMES:
Complication | From date of treatment until the date of first documented complication, assessed up to 24 months
  Complications included hoarseness, infection, hematoma, airway obstruction, and permanent hypoparathyroidism.

CONTACTS AND LOCATIONS:
Locations (1):
- ChinaPLAGH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Some of the data generated or analyzed during the study are available from the corresponding author by reasonable request.